CLINICAL TRIAL: NCT00539370
Title: Laboratory of Immunology/National Eye Institute Repository
Brief Title: Human Samples and Data Repository
Status: Terminated | Type: Observational
Why Stopped: The investigator is no longer employed at NIH.
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070213; 07-EI-0213
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Uveitis; Scleritis
Keywords: Scleritis; Intermediate Uveitis; Posterior Uveitis; Intraocular Inflammatory Disease; Data Analysis; Data Collection; Sample Analysis
MeSH Terms: conditions — Uveitis; Scleritis; Uveitis, Intermediate; Uveitis, Posterior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, DNA, and pharmacokinetic samples have been retained

SUMMARY:
This protocol will enable IRB (institutional review board) review of proposed research using human samples and data collected under the terminated NIH studies 04-EI-0065 and 96-EI-0096. Data and samples may include demographic and personal health information, psychological or psychiatric testing, blood, urine, CSF or other body fluids or tissues and results of medical and physiological evaluation and medical imaging.

Data and sample analyses are limited to those approved under the original protocols unless additional specific institutional review board approval is obtained.

DETAILED DESCRIPTION:
Objective: This protocol will enable prospective IRB review of research using human samples and data collected under other branch protocols.

Study population: Participants that were followed in terminated branch protocols under which data or samples were collected.

Design: Samples and data will be brought under this protocol, analyzed and stored for uses specified in the original protocols and as additionally approved by the IRB.

Outcome: The outcome of this protocol will be the storage, tracking, and utilization of samples and data obtained under terminated protocols.

Purpose: The purpose of this protocol is to enable prospective IRB review of research using human samples and data collected under other branch protocols.

Participants: Participants who previously participated in NIH protocols whose wishes regarding use of their samples or data for research other than that specified in the initial protocol is not known may be enrolled in this protocol. At this time, there are no additional analyses planned outside of the original protocols, apart from those listed below. Participant consent or IRB approval for a waiver of additional informed consent will be sought prior to initiation of additional analyses.

ELIGIBILITY:
* Data Analysis Study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who were followed in terminated branch protocols under which data or samples were collected.
Sampling Method: Non-Probability Sample
Enrollment: 1862 (Actual)
Dates: Start 2007-08-29 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2022-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-EI-0213.html